CLINICAL TRIAL: NCT02439385
Title: First Line Avastin/FOLFIRI in Combination With Curcumin-containing Supplement in Colorectal Cancer Patients With Unresectable Metastasis
Brief Title: Avastin/FOLFIRI in Combination With Curcumin in Colorectal Cancer Patients With Unresectable Metastasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Collaborators: Aju Pharm (Unknown)
Responsible Party: Principal Investigator, Jeong-Heum Baek, MD, Professor, Gachon University Gil Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAIRB2015-87
Record Dates: First submitted 2015-05-02; First posted 2015-05-08 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Cancer
Keywords: Curcumin; Avastin; FOLFIRI; Colorectal cancer; Unresectable metastasis
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Avastin/FOLFIRI with curcumin (Experimental): Patients will receive first line Avastin/FOLFIRI in combination with curcumin-containing supplement
  Interventions: Drug: Avastin/FOLFIRI; Dietary Supplement: Curcumin

INTERVENTIONS:
Drug: Avastin/FOLFIRI — Avastin: 5mg/kg iv on day1, every 14 days. Irinotecan: 180 mg /m2 iv on day1, every 14 days. Leucovorin: 200 mg/m2 iv on day1,2 every 14 days. 5-fluorouracil bolus: 400 mg/m2 iv on day1,2 every 14 days. 5-fluorouracil infusion: 1200 mg/m2 iv on day1,2 every 14 days.
  Other Names: Bevacizumab/FOLFIRI
Dietary Supplement: Curcumin — Dietary supplement of nanostructured lipid curcumin particle 100mg po bid daily

SUMMARY:
Oral curcumin-containing supplement will be given to colorectal cancer patients with unresectable metastases who will be starting Avastin/FOLFIRI chemotherapy for up to completion of (or withdrawal from) chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age : 20 Years and older
* Histologically confirmed adenocarcinoma of the colon or rectum
* Patients with primary colon or rectal cancer and unresectable metastatic lesions.
* Patients with no primary cancer related symptoms.
* ECOG performance status of 0 - 2
* Appropriate organ functions (hepatic transaminases - less than 5 times the normal range; bilirubin - less than 2 times the normal range; creatinine serum - less than 1.5 times the normal range; thrombocyte - more than 100,000/µl; neutrophil - more than 1,500/µl)
* ASA score of < 3
* An informed consent form has been signed by the patient.

Exclusion Criteria:

* Colorectal cancer other than adenocarcinoma
* The patient received adjuvant chemotherapy within the past 6 months.
* The patient received chemotherapy for metastatic colon cancer.
* The patient was planning to have curative surgery for the metastatic lesions.
* Patients with peritoneal carcinomatosis.
* Patients with primary tumor related complications such as intestinal obstruction, intractable bleeding, and perforation, that needs to be treated.
* ASA score of > 4
* The patient has chronic hepatitis or cirrhosis. An asymptomatic HBV or HCV carrier can participate.
* Patients with an active infection, which need antibiotic therapy, during the randomization period.
* Pregnant or breastfeeding women
* Patients with another different malignant tumor during the past 5 years. Patients with treated non-melanoma skin cancer or cervical cancer can be enrolled in this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-08-24 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  The primary end point of this study is to evaluate progression-free survival in colorectal cancer patients with unresectable metastasis after treatment with first line Avastin/FOLFIRI in combination with a dietary supplement of nanostructured lipid curcumin particle (Aju Pharm, Korea), which improved biotransformation and bioavailability profiles of curcumin.

SECONDARY OUTCOMES:
Overall survival rate | 3 years
  Overall survival will be measured in months. Overall survival will be measured in months. Overall survival will be measured in months. Overall survival will be measured in months.
Overall response rate | 2 years
  According to RECIST criteria v1.1
Safety (assessed by toxicity grades defined by NCI-CTCAE (version 4.0) | 2 years
  Safety as assessed by toxicity grades defined by NCI-CTCAE (version 4.0)
Quality of life (QoL) | 2 years
  QoL measured by the FACT-G (version 4, Korean version)
Fatigue (FACIT-Fatigue scale (version 4, Korean version) | 2 years
  Fatigue measured by the FACIT-Fatigue scale (version 4, Korean version)

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Heum Baek, MD, Ph.D, Principal Investigator — Gachon University Gil Medical Center

REFERENCES:
- [Derived] Jeon Y, Sym SJ, Yoo BK, Baek JH. Long-term Survival, Tolerability, and Safety of First-Line Bevacizumab and FOLFIRI in Combination With Ginsenoside-Modified Nanostructured Lipid Carrier Containing Curcumin in Patients With Unresectable Metastatic Colorectal Cancer. Integr Cancer Ther. 2022 Jan-Dec;21:15347354221105498. doi: 10.1177/15347354221105498. PMID 35695002